CLINICAL TRIAL: NCT02004951
Title: BATTLE Trial: Bare Metal Stent Versus Paclitaxel Eluting Stent in the Setting of Primary Stenting of Intermediate Length Femoropopliteal Lesions
Acronym: BATTLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Batch recall for Misago Terumo self-expanding peripheral stent systems.(withdrawal from the market)
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC13_0290
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Peripheral Arterial Disease; Femoropopliteal Lesions
Keywords: Superficial femoral artery; paclitaxel; stent; self expandable; restenosis; endovascular; above-the-knee intermediate length
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misago RX (Misago RX, Terumo Corp., Tokyo (Other): The Misago RX is a peripheral stent (Misago RX, Terumo Corp., Tokyo, Japan) indicated to treat iliac and femoropopliteal arteries. The Misago RX is a flexible self-expanding nitinol stent that is delivered via a RX monorail delivery catheter.
  Interventions: Device: Misago RX
- Zilver PTX (Cook Medical, Bloomington, IN, USA) (Other): Zilver PTX (Cook Medical, Bloomington, IN, USA) is a nitinol stent with a polymer-free paclitaxel coating designed to treat the above- the-knee femoropopliteal arteries. The anti-proliferative drug is the paclitaxel, a cytotoxic drug. The Zilver PTX stent is delivered via a over-the-wire system.
  Interventions: Device: Zilver PTX

INTERVENTIONS:
Device: Misago RX
  Other Names: Treatment of above-the-knee intermediate length femoropopliteal lesions
  Arms: Misago RX (Misago RX, Terumo Corp., Tokyo
Device: Zilver PTX
  Arms: Zilver PTX (Cook Medical, Bloomington, IN, USA)

SUMMARY:
Over the past years, endovascular interventions have become an important part of treatment in patients with peripheral arterial disease.1 Indication for endovascular repair of femoropopliteal lesions has been considerably enlarged as shown in the TASC classification.1 Enlargement of endovascular therapy indication was based on patient choice for a less invasive technique and evidence based medicine. Consequently, TASC classification of lesions has been modified to reflect increased evidence for endovascular treatment of more extensive femoropopliteal lesions, and indication for endovascular repair has been enlarged to more severe TASC types. In summary, endovascular treatment is indicated for TASC A and B lesions which correspond to femoropopliteal lesions ≤15-cm. To treat these lesions, the interventionalists have at their disposal a huge tool box. Evaluation of these tools is crucial to determine the right treatment strategy to avoid further reinterventions and overcosts.

The objective of the BATTLE trial is to compare a bare metal self expandable nitinol stent (Misago RX) versus a paclitaxel eluting stent (Zilver PTX) in the treatment of above-the-knee intermediate length femoropopliteal lesions.

From hospitals in Europe (France, Switzerland) we will randomly assign patients with symptomatic atherosclerotic femoropopliteal lesions to be treated either by bare metal stent or paclitaxel eluting stent. In total, 186 patients will be randomized (93 per group).

ELIGIBILITY:
Inclusion criteria

* Patient ≥18 years
* Patient has a history of symptomatic peripheral arterial disease (Rutherford classification: 2-5)
* Lesion is eligible for treatment with a maximum of 2 stents per lesion (treatment of both legs is not permitted)
* Patient is affiliated to the Social Security or equivalent system
* Patient has been informed of the nature of the study, agrees to its provisions (and only for swiss centers, has signed the informed consent form prior to any study related procedure)
* Patient agrees to undergo all protocol required follow-up examinations and requirements at the investigational site
* Reference vessel diameter 4 to 7-mm determined by CT scan (RVD obtained from averaging 5-mm segments proximal and distal to the lesions)
* Target lesion has a pre-procedure percent diameter stenosis of ≥ 50% DS
* De novo atherosclerotic lesions (stenosis and/or occlusion) of the superficial femoral artery, the proximal popliteal artery (P1), or both. The treatment area in the SFA and popliteal artery extended from 1 cm below the origin of the profunda femoris artery to 3 cm above the proximal margin of the intercondylar fossa of the femur.
* Target lesion (single or multiple) has a maximal total length =14-cm and a minimal length = 2-cm
* At least 1 patent runoff vessel (<50% DS throughout its course). The inflow artery(ies) cannot be treated using a drug eluting stent or drug coated balloon.

Exclusion Criteria

* Asymptomatic lesion
* Restenosis
* No atheromatous disease
* Untreated >50% DS of the inflow tract
* Resting ankle brachial index (ABI) unavailable
* Female of child bearing potential
* Patient has received, or is on the waiting list for a major organ transplant
* Patient has a history of coagulopathy or will refuse blood transfusions
* Patient is receiving or scheduled to receive anticancer therapy for malignancy within 1 year prior to or after the procedure
* Severe concomitant disease with life expectation < one year
* Known allergy to paclitaxel
* Contraindication to Aspirin or Clopidogrel and Ticlopidin (the patient must be able to receive Dual Anti-Platelet Treatment for 2 months after the procedure)
* Patient has an infected wound or osteomyelitis on the ipsilateral extremity or foot.
* Patient has had prior major amputation to the ipsilateral (target) extremity
* Patient is not able to give informed consent (and only for swiss centers)
* Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints Note: Trials requiring extended follow-up for products that were investigational, but have become commercially available since then, are not considered investigational trials
* Patient has previously had, or requires, bypass surgery, endarterectomy or other vascular surgery on any vessel of the ipsilateral extremity
* In the Investigator's opinion patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
* Target lesion lies within or adjacent to an aneurysm
* Patient with an allergy to contrast agent
* Patient with a severe allergy to metal
* Surgery or endovascular intervention of the target member within 14 days preceding the BATTLE procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Freedom from in-stent restenosis at 1 year | 1 year
  It was defined by restenosis of >50% and by a peak systolic velocity index >2.4 at the target lesion.

SECONDARY OUTCOMES:
residual diameter stenosis | Day 0
  Technical success defined achievement of a final residual diameter stenosis of <30% on the procedural completion angiogram.
Primary sustained clinical improvement | 1 month, 12 months and 24 months
  sustained upward shift of _1 category of the Rutherford classification for claudicants and by wound healing and rest pain resolution for patients in CLI, without the need for repeated TLR in surviving patients.
Secondary sustained clinical improvement | 1 month, 12 months and 24 months
  primary sustained clinical improvement including the need for repeated TLR.
Primary patency | 1 month, 12 months and 24 months
  patency without any percutaneous or surgical intervention in the treated segment or in the adjacent areas.
Major adverse events | 1 month, 12 months and 24 months
  MACEs including all deaths, major amputation.
Limb salvage | 1 month, 12 months and 24 months
  freedom from major ipsilateral amputations
Death | 1 month, 12 months and 24 months
  Death (all cause)
Ankle brachial index | 1 month, 6 months, 12 months and 24 months
  Ankle brachial index
Target Extremity Revascularization (TER) | 1 month, 12 months and 24 months
  TER is defined as any percutaneous intervention or surgical bypass of any segment of the target extremity. The target extremity is defined as the ipsilateral limb arteries proximal and distal to the target lesion, which includes upstream and downstream branches and excludes the target lesion itself.
Target lesion revascularization (TLR) | 1 month, 12 months and 24 months
  TLR expresses the frequency of the need for repeated procedures (endovascular or surgical) due to a problem arising from the stent (1 cm proximally and distally to include edge phenomena) in surviving patients with preserved limb.
Stent fracture | 1 month, 12 months and 24 months
  Stent fractures were assessed by biplane x-rays
EQ-5D-3L questionnaire | 1 month, 12 months and 24 months
  Quality of life - EQ-5D-3L questionnaire EQ-5D-3L = European Quality of Life 5 Dimensions and 3 Lines Scale from 0 to 100. 0 =Worst imaginable state of health 100= Best imaginable state of health
Economic analysis objective | 2 years
  Incremental cost-effectiveness ratio (ICER) based on quality of life for CUA and on freedom from in-stent restenosis for CEA

CONTACTS AND LOCATIONS:
Overall Officials: Yann GOUEFFIC, Professor, Study Chair — Nantes University Hospital
Locations (11):
- France (11):
  - Clinique d'Antony, Antony
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Pierre Oudot Bourgoin Jallieu, Bourgoin
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - AP-HP, Hôpital Henri Mondor, Créteil
  - CHU de Lyon, Lyon
  - CHU Nantes, Nantes
  - Clinique Ollioules, Ollioules
  - CHU de Rennes, Rennes
  - Clinique Pasteur, Toulouse

REFERENCES:
- [Derived] Goueffic Y, Kaladji A, Guyomarch B, Montagne C, Fairier D, Gestin S, Riche VP, Vent PA, Chaillou P, Costargent A, Patra P. Bare metal stent versus paclitaxel eluting stent for intermediate length femoropopliteal arterial lesions (BATTLE trial): study protocol for a randomized controlled trial. Trials. 2014 Oct 30;15:423. doi: 10.1186/1745-6215-15-423. PMID 25359394